CLINICAL TRIAL: NCT03742102
Title: A Phase IB/II, 2-stage, Open-label, Multicenter Study to Determine the Efficacy and Safety of Durvalumab (MEDI4736) + Paclitaxel and Durvalumab (MEDI4736) in Combination With Novel Oncology Therapies With or Without Paclitaxel for First-line Metastatic Triple Negative Breast Cancer
Brief Title: A Study of Novel Anti-cancer Agents in Patients With Metastatic Triple Negative Breast Cancer
Acronym: BEGONIA
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D933LC00001; 2018-000764-29 (EudraCT Number)
Record Dates: First submitted 2018-10-25; First posted 2018-11-15 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Triple Negative Breast Neoplasms
Keywords: Breast Cancer; TNBC; Triple Negative; Triple Negative Breast Cancer; Triple-Negative Breast Cancer; Triple-Negative Breast Neoplasm; ER-Negative PR-Negative HER2-Negative Breast Cancer; ER-Negative PR-Negative HER2-Negative Breast Neoplasms; PD-L1 high TNBC
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — durvalumab; capivasertib; Paclitaxel; trastuzumab deruxtecan

STUDY DESIGN:
Intervention Model Description: Part 1:
  At least 20 patients in the durvalumab-paclitaxel arm and at least 30 patients in each of the other novel treatment combination arms will be enrolled, for a total of approximately 140 patients (durvalumab + paclitaxel arm and 4 novel treatment combination arms). Additional patients may be enrolled in order to have 20 or 30 evaluable (i.e. dosed) patients per durvalumab - paclitaxel arm or novel treatment combination arm, respectively.
  Part 2:
  Approximately 27 patients will be assigned to each treatment arm, for an anticipated total of 57 response-evaluable patients per arm (ie, 30 patients in Part 1 and 27 patients in Part 2 per treatment arm, with the exception of Arm 1, which will enroll 20 patients in Part 1 and will not be expanded to Part 2). Patient expansion from 30 patients in Part 1 to an additional 27 patients from Part 2 will be determined based on a futility analysis utilizing a Simon 2 Stage design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1 (Experimental): durvalumab + paclitaxel
  Interventions: Drug: Durvalumab; Drug: Paclitaxel
- Arm 2 (Experimental): durvalumab + paclitaxel + capivasertib
  Interventions: Drug: Durvalumab; Drug: Capivasertib; Drug: Paclitaxel
- Arm 5 (Experimental): durvalumab + paclitaxel + oleclumab
  Interventions: Drug: Durvalumab; Drug: Oleclumab; Drug: Paclitaxel
- Arm 6 (Experimental): durvalumab + trastuzumab deruxtecan
  Interventions: Drug: Durvalumab; Drug: Trastuzumab deruxtecan
- Arm 7 (Experimental): durvalumab + datopotamab deruxtecan
  Interventions: Drug: Durvalumab; Drug: Datopotamab deruxtecan
- Arm 8 (Experimental): durvalumab + datopotomab deruxtecan (patients with PD-L1 positive status)
  Interventions: Drug: Durvalumab; Drug: Datopotamab deruxtecan

INTERVENTIONS:
Drug: Durvalumab — Durvalumab iv Every 4 weeks (q4w) or 3 weeks (q3w) Arm 6, 7 and 8
  Other Names: MEDI4736
Drug: Capivasertib — Capivasertib oral bid 4-week cycles; 3 weeks on (dosing on days 2,3,4 and 5) and 1 week off
  Other Names: AZD5363
  Arms: Arm 2
Drug: Oleclumab — Oleclumab iv Every 2 weeks (q2w) for first 2 cycles (days 1 and 15 in cycles 1 and 2), then every 4 weeks (q4w) starting at cycle 3 day 1
  Other Names: MEDI9447
  Arms: Arm 5
Drug: Paclitaxel — Paclitaxel iv 4-week cycles: 3 weeks once weekly (q1w) and 1 week off
  Arms: Arm 1; Arm 2; Arm 5
Drug: Trastuzumab deruxtecan — Trastuzumab deruxtecan iv 3-week cycles (once weekly) q3w
  Other Names: DS-8201a
  Arms: Arm 6
Drug: Datopotamab deruxtecan — Datopotamab deruxtecan iv 3-week cycles (once weekly) q3w
  Other Names: Dato-DXd; DS-1062a
  Arms: Arm 7; Arm 8

SUMMARY:
This study is designed to determine the efficacy and safety of durvalumab in combination with novel oncology therapies with or without paclitaxel and durvalumab + paclitaxel for first-line metastatic triple negative breast cancer

DETAILED DESCRIPTION:
This is a Phase IB/II, 2-stage, open-label, multicenter study to determine the efficacy and safety of durvalumab in combination with novel oncology therapies (i.e. therapies designed for immune modulation) with or without paclitaxel and durvalumab + paclitaxel as first-line treatment in patients with metastatic triple negative breast cancer (TNBC). The study is designed to concurrently evaluate potential novel treatment combinations with clinical promise using a 2-stage approach. The study will use a Simon 2-Stage design to evaluate which cohorts may proceed to expansion.

Part 1 is a Phase IB study of safety and initial efficacy, and Part 2 may expand patient enrollment if adequate efficacy signal is observed in Part 1. The treatment regimens evaluated in Part 2 will depend on the evaluation of safety and efficacy outcomes in Part 1.

ELIGIBILITY:
Inclusion criteria

1. Female
2. At least 18 years of age at the time of screening
3. Patient must have locally confirmed advanced/unresectable or metastatic TNBC.
4. No prior treatment for metastatic (Stage IV) TNBC
5. Patient must have at least 1 lesion, not previously irradiated, that can be accurately measured
6. WHO/ECOG status at 0 or 1 at enrollment

Patients enrolled to Arm 6 (durvalumab and DS-8201a) Must provide documentation of locally determined advanced/unresectable or metastatic TNBC with HER2 low tumor expression (IHC 2+/ISH-, IHC 1+/ISH-, or IHC 1+/ISH untested)

Patients enrolled in Arm 8 (durvalumab + Dato-DXd) Must have PD-L1 positive tumor as determined by an IHC based assay

Exclusion criteria

1. History of allogeneic organ transplantation
2. Active or prior documented autoimmune or inflammatory disorders
3. Active infection including tuberculosis, hepatitis B (known positive HBV surface antigen [HBsAg] result), hepatitis C virus (HCV), or human immunodeficiency virus (positive HIV 1/2 antibodies)
4. Untreated CNS metastases
5. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
6. Any concurrent chemotherapy, IP, or biologic therapy for cancer treatment
7. Female patients who are pregnant, breastfeeding
8. Cardiac Ejection Fraction less than 50%

Patients enrolled in Arm 2 only:

1. Potent inhibitors or inducers or substrates of CYP3A4 or substrates of CYP2C9 or CYP2D6 within 2 weeks before the first dose of study treatment (3 weeks for St John's Wort)
2. Diagnosis of diabetes mellitus Type I or diabetes mellitus Type II requiring insulin treatment.
3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure, hypokalemia, potential for torsades de pointes, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age, or any concomitant medication known to prolong the QT interval
4. Prior treatment with PI3K inhibitors, AKT inhibitors, or mammalian target of rapamycin (mTOR) inhibitors.

Patients enrolled in Arm 5 only: History of venous thromboembolism in the past 3 months

Patients enrolled in Arm 7 and 8 only: Clinically significant corneal disease in the opinion of the Investigator.

Patients enrolled in Arm 6, 7 and 8 only:

1. History of or active interstitial lung disease/pneumonitis
2. Use of chloroquine or hydroxychloroquine in <14 days prior to Day 1 of DS-8201a (Arm 6) or Dato-DXd (DS-1062a; Arm 7 and 8) treatment
3. Patients enrolled in Arm 6 only: Previously been diagnosed as HER2+ or received HER2-targeted therapy.

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 243 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2027-02-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid, MD, PhD, Principal Investigator — Barts Cancer Institute
Locations (27):
- United States (7):
  - Research Site, Tucson, Arizona
  - Research Site, Columbia, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Grand Rapids, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Dallas, Texas
  - Research Site, Williamsburg, Virginia
- Canada (4):
  - Research Site, Kelowna, British Columbia
  - Research Site, London, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
- Poland (6):
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Opole
  - Research Site, Rzeszów
  - Research Site, Warsaw
- Research Site, Seoul, South Korea
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Breast Cancer Study Locator details (for US) — https://www.breastcancerstudylocator.com/trial/listing/188918
- See also: Study Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933LC00001&attachmentIdentifier=56218ffb-f5f4-4869-8215-7f6c6c2b5bab&fileName=D933LC00001_CSP.pdf&versionIdentifier=
- See also: SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933LC00001&attachmentIdentifier=ce6580e5-178a-4bce-9659-c5b4e8a7a03e&fileName=d933lc00001-sap.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D933LC00001&attachmentIdentifier=71aaba78-8436-413e-81a1-d6cbf5d41056&fileName=d933lc00001-study-synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data cut-off is 30Jun23 for Arms 1,2,5,6 and 29Nov24 for Arms 7-8
Pre-assignment Details: Part 1 evaluated safety (with safety run-in Arms 2, 5, 6 and 7), efficacy, PK and immunogenicity for durvalumab combinations. Enrolment was expanded in Part 2, if pre-defined Part 1 efficacy signals were observed.
  Per the CSP and SAP, participants from Part 1 and 2 were analyzed together, no separate analyses by Part are available.
  Arms including Part 1 only: 1, 2, 5, 8.
  Arms including Part 1 and 2: Arms 6 and 7. No expansion to Part 2 was planned for Arm 8.
Groups:
- Arm 1: Durvalumab 1500 mg q4w, IV + Paclitaxel 90 mg/m2, IV, q4w: 3 weeks on (D1, D8, and D15) and 1 week off
- Arm 2: Durvalumab 1500 mg q4w, IV + Paclitaxel 80 mg/m2 or 90 mg/m2, IV, q4w: 3 weeks on (D1, D8, and D15) and 1 week off+ Capivasertib 400 mg, oral use bid 4 days on (D2, D3, D4, and D5) and 3 days off 4-week cycles: 3 weeks on (D1, D8, and D15) and 1 week off
- Arm 5: Durvalumab 1500 mg q4w, IV + Paclitaxel 90 mg/m2, IV, q4w: 3 weeks on (D1, D8, and D15) and 1 week off + Oleclumab 3000 mg q2w for first 2 cycles, IV (D1 and D15 of C1 and C2), then q4w starting at C3 (D1)
- Arm 6: Durvalumab 1120 mg q3w, IV + Trastuzumab Deruxtecan 5.4 mg/kg q3w, IV
- Arm 7: Durvalumab 1120 mg q3w, IV + Datopotamab Deruxtecan 6.0 mg/kg q3w, IV
- Arm 8: Durvalumab 1120 mg q3w, IV + Datopotomab Deruxtecan 6.0 mg/kg q3w, IV (patients with PD-L1 positive status)
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 5 | Arm 6 | Arm 7 | Arm 8
Started (Received study treatment) | 23 | 31 | 33 | 58 | 62 | 33
Completed (All patients in Arms 1, 2, 5 and 6 that were ongoing at the time of DCO (30Jun2023) were not expected to have a status of 'Completed'.) | 0 | 0 | 0 | 0 | 6 | 3
Not Completed | 23 | 31 | 33 | 58 | 56 | 30
Not completed — Death | 14 | 17 | 25 | 22 | 28 | 3
Not completed — Ongoing study at time of data cut-off (30Jun23 for Arms 1-6 and 29Nov24 for Arms 7-8) | 8 | 9 | 5 | 33 | 24 | 25
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 3 | 2 | 3 | 2
Not completed — Reason unknown | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 5 | Arm 6 | Arm 7 | Arm 8 | Total
Number analyzed (Participants) | 23 | 31 | 33 | 58 | 62 | 33 | 240
Age, Continuous [Median (Full Range); unit: Years] | 52 [30 to 62] | 51 [32 to 71] | 54 [33 to 72] | 54 [29 to 81] | 53 [31 to 74] | 47 [29 to 74] | 52 [29 to 81]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 23 | 31 | 33 | 58 | 62 | 33 | 240
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 23 | 31 | 33 | 56 | 62 | 33 | 238
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 0 | 1 | 2 | 4 | 1 | 8
  Asian | 17 | 16 | 17 | 16 | 15 | 20 | 101
  White | 5 | 15 | 15 | 39 | 39 | 11 | 124
  Other | 1 | 0 | 0 | 1 | 4 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT) Events
Description: The occurrence of a severe adverse event (meeting pre-specified criteria) that is at least possibly related to durvalumab and/or the novel oncology therapy in 6 DLT-evaluable patients
Time Frame: From the time of first dose until completion of the first cycle (28 days for Arms 2-5, 21 days for Arms 6-7 (no safety run-in for Arms 1 and 8))
Population: Safety analysis set
Measure: Number; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 5 | Arm 6 | Arm 7 | Arm 8
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 0
Participants |  | 0 | 0 | 0 | 0 |

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Percentage of evaluable patients with a confirmed Investigator-assessed response of CR (complete response) or PR (partial response). Confirmed response is defined as at least one visit response of CR or PR confirmed by a follow-up scan at least 4 weeks later showing CR or PR.
Time Frame: Tumor assessments: every 8 wks (Arms 1-5) or every 6 wks (Arms 6-8) until wk 48, then every 12 wks from first IP dose until radiologic progression, death, withdrawal of consent, or study completion; up to max 54 mos (observed longest duration in Arm 1)
Population: Number of patients with measurable disease at baseline who have had the opportunity to complete at least 2 on-treatment disease assessments
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm 1 | Arm 2 | Arm 5 | Arm 6 | Arm 7 | Arm 8
Number analyzed (Participants) | 23 | 31 | 33 | 58 | 62 | 33
Percentage of patients | 56.5 [34.5 to 76.8] | 54.8 [36.0 to 72.7] | 51.5 [33.5 to 69.2] | 62.1 [48.4 to 74.5] | 79.0 [66.8 to 88.3] | 81.8 [64.5 to 93.0]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Time from date of first dose (at least one study intervention [durvalumab, paclitxel or novel oncology therapy]) until the date of objective radiological disease progression using RECIST 1.1 or death (by any cause in the absence of progression)
Time Frame: as for outcome 2
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1 | Arm 2 | Arm 5 | Arm 6 | Arm 7 | Arm 8
Number analyzed (Participants) | 23 | 31 | 33 | 58 | 62 | 33
Months | 7.3 [5.4 to 11.3] | 6.4 [5.4 to 10.3] | 8.3 [4.8 to 9.3] | 12.6 [8.4 to 16.3] | 14.0 [11.0 to 21.1] | 11.2 [6.9 to 13.8]

4. Secondary Outcome: Duration of Response (DoR)
Description: Time from the date of first documented response (which is subsequently confirmed) until the first date of documented progression (PD) or death in the absence of PD (ie, date of PFS event or censoring - date of first response + 1). If a patient does not progress following a response, then their DoR will be censored at the last evaluable disease assessment date
Time Frame: as for outcome 2
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1 | Arm 2 | Arm 5 | Arm 6 | Arm 7 | Arm 8
Number analyzed (Participants) | 23 | 31 | 33 | 58 | 62 | 33
Months | 5.6 [3.75 to 26.12] | 7.9 [3.98 to 14.59] | 7.8 [5.42 to 17.77] | 15.2 [8.44 to NA] — NA - Not calculable due to insufficient number of events for upper limit of confidence interval | 17.6 [10.51 to 27.27] | 11.5 [5.16 to NA] — NA - Not calculable due to insufficient number of events for upper limit of confidence interval

5. Secondary Outcome: Overall Survival (Count)
Description: Number of patients with overall survival, the time from date of first dose (at least one study intervention [durvalumab, paclitxel or novel oncology therapy]) until the date of death by any cause
Time Frame: From date of first dose until date of death due to any cause; up to the maximum of 54 months (observed longest duration in Arm 1)
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 5 | Arm 6 | Arm 7 | Arm 8
Number analyzed (Participants) | 23 | 31 | 33 | 58 | 62 | 33
Participants
  Died | 14 | 18 | 25 | 22 | 28 | 3
  Alive at data cut-off | 8 | 9 | 5 | 33 | 30 | 28
  Terminated prior to death | 1 | 4 | 3 | 3 | 4 | 2

6. Secondary Outcome: Overall Survival (Duration)
Description: Time from date of first dose (at least one study intervention [durvalumab, paclitxel or novel oncology therapy]) until the date of death by any cause
Time Frame: From date of first dose of IP until date of death due to any cause; up to the maximum of 54 months (observed longest duration in Arm 1)
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1 | Arm 2 | Arm 5 | Arm 6 | Arm 7 | Arm 8
Number analyzed (Participants) | 23 | 31 | 33 | 58 | 62 | 33
Months | 30.0 [13.0 to NA] — NA - Not calculable due to insufficient number of events for upper limit of confidence interval | 32.6 [12.9 to 40.0] | 24.8 [18.6 to 31.9] | 30.3 [18.8 to NA] — NA - Not calculable due to insufficient number of events for upper limit of confidence interval | NA [23.2 to NA] — NA - Not calculable due to insufficient number of events for upper limit of confidence interval | NA [NA to NA] — NA - Not calculable due to insufficient number of events for upper limit of confidence interval

7. Secondary Outcome: Progression-free Survival at 6 Months (PFS6)
Description: Percentage of patients alive and progression-free at 6 months following date of first dose (at least one study intervention [durvalumab, paclitxel or novel oncology therapy])
Time Frame: 6 months following date of first dose
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1 | Arm 2 | Arm 5 | Arm 6 | Arm 7 | Arm 8
Number analyzed (Participants) | 23 | 31 | 33 | 58 | 62 | 33
Percentage of participants | 56.5 [34.3 to 73.8] | 52.4 [33.1 to 68.5] | 65.3 [46.0 to 79.1] | 75.2 [61.8 to 84.5] | 79.8 [67.2 to 88.0] | 78.2 [59.5 to 89.0]

ADVERSE EVENTS:
Time Frame: From the time of signature of informed consent up to 90 days after the last dose of study treatment. If an event starts post this period noted and is considered to be due to a late-onset toxicity to study drug, then it should be reported as an AE/SAE. Maximum duration of approximately 54 months.
Description: Arms 1-6 used MedDRA 26.0; Arms 7-8 used MedDRA 27.1
Groups:
- Durva + Pac; Durva + Pac + Capi 400mg Bid; Durva + Pac + Olec 3000mg; Durva + DS-8201a; Durva + Dato-DXd; Durva + Dato-DXd (PD-L1 High): Description (Arm-group)
Arm/Group | Durva + Pac | Durva + Pac + Capi 400mg Bid | Durva + Pac + Olec 3000mg | Durva + DS-8201a | Durva + Dato-DXd | Durva + Dato-DXd (PD-L1 High)
All-Cause Mortality (participants affected / at risk) | 14/23 | 18/31 | 25/33 | 22/58 | 28/62 | 3/33
Serious Adverse Events (participants affected / at risk) | 1/23 | 11/31 | 4/33 | 16/58 | 18/62 | 5/33
Other Adverse Events (participants affected / at risk) | 22/23 | 30/31 | 32/33 | 57/58 | 62/62 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durva + Pac (N=23) | Durva + Pac + Capi 400mg Bid (N=31) | Durva + Pac + Olec 3000mg (N=33) | Durva + DS-8201a (N=58) | Durva + Dato-DXd (N=62) | Durva + Dato-DXd (PD-L1 High) (N=33)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flap necrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiation necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic enzymes increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durva + Pac (N=23) | Durva + Pac + Capi 400mg Bid (N=31) | Durva + Pac + Olec 3000mg (N=33) | Durva + DS-8201a (N=58) | Durva + Dato-DXd (N=62) | Durva + Dato-DXd (PD-L1 High) (N=33)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0) | 8 (20) | 4 (4) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (4) | 1 (2) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 4 (4) | 7 (9) | 13 (16) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 3 (4) | 9 (11) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 2 (2) | 6 (6) | 4 (4) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (15) | 3 (3) | 8 (12) | 4 (4) | 2 (6) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 4 (5) | 0 (0)
Dizziness (Nervous system disorders) | 4 (6) | 2 (2) | 5 (5) | 4 (4) | 8 (14) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 2 (5) | 5 (8) | 12 (13) | 9 (9) | 9 (17) | 3 (6)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 6 (6) | 8 (9) | 1 (1) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 4 (8) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 13 (14) | 7 (7) | 13 (13) | 2 (2) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 5 (6) | 3 (3) | 5 (5) | 7 (8) | 4 (4)
Hypothyroidism (Endocrine disorders) | 6 (6) | 1 (1) | 7 (7) | 15 (16) | 11 (11) | 8 (8)
Dysuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (2) | 2 (2) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 7 (7) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 8 (10) | 7 (7) | 6 (8) | 12 (13) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 3 (3) | 4 (4) | 5 (5) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 7 (9) | 5 (5)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 17 (17) | 4 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 2 (2) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (14) | 11 (11) | 16 (16) | 16 (16) | 31 (33) | 13 (14)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 11 (11) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 4 (4) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Onycholysis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 10 (12) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (9) | 10 (11) | 6 (7) | 3 (6) | 10 (12) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 9 (12) | 18 (27) | 9 (11) | 7 (9) | 21 (30) | 13 (17)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (6) | 1 (2) | 1 (1) | 4 (5) | 3 (5)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 7 (8) | 5 (6)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 2 (3) | 2 (4) | 4 (4) | 4 (4) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (12) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 2 (2)
Limbal stem cell deficiency (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Punctate keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 5 (6)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 7 (11) | 4 (6) | 16 (23) | 9 (10) | 3 (5)
Visual impairment (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 3 (3) | 3 (3) | 4 (4) | 6 (7) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 6 (6) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (6) | 2 (2) | 5 (5) | 20 (26) | 31 (36) | 10 (12)
Diarrhoea (Gastrointestinal disorders) | 3 (7) | 21 (42) | 11 (15) | 13 (22) | 10 (26) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 6 (6) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (10) | 1 (1) | 3 (3) | 8 (9) | 6 (6) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (2) | 4 (4) | 2 (3) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 4 (4) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (27) | 8 (11) | 11 (17) | 46 (71) | 42 (81) | 18 (30)
Stomatitis (Gastrointestinal disorders) | 4 (5) | 4 (5) | 6 (6) | 9 (11) | 43 (88) | 27 (35)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (6) | 3 (4) | 2 (2) | 18 (24) | 18 (42) | 9 (12)
Asthenia (General disorders) | 4 (6) | 2 (2) | 4 (5) | 12 (16) | 7 (9) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 9 (13) | 10 (12) | 6 (6) | 31 (36) | 30 (46) | 12 (13)
Generalised oedema (General disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Oedema peripheral (General disorders) | 7 (7) | 1 (2) | 6 (6) | 4 (4) | 4 (5) | 0 (0)
Pyrexia (General disorders) | 4 (8) | 8 (15) | 2 (2) | 8 (15) | 5 (6) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 8 (29) | 0 (0) | 19 (46) | 3 (3) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Covid-19 (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 11 (12) | 15 (18) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 9 (19) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (4) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 4 (5) | 3 (4)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (5) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 2 (5) | 4 (6) | 8 (10) | 8 (16) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3) | 5 (6) | 2 (2) | 3 (5) | 10 (16) | 1 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 6 (17) | 4 (5)
Alanine aminotransferase increased (Investigations) | 5 (5) | 5 (6) | 2 (2) | 13 (17) | 7 (9) | 6 (7)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 12 (25) | 8 (11)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 5 (6) | 2 (2) | 12 (17) | 7 (9) | 4 (6)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 4 (7) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (10) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (2) | 2 (2) | 6 (13) | 4 (7) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 4 (6) | 2 (2) | 1 (1)
Lipase increased (Investigations) | 2 (3) | 0 (0) | 3 (3) | 5 (7) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 7 (28) | 4 (10) | 2 (3) | 1 (3) | 1 (1) | 2 (3)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 6 (7) | 1 (2)
White blood cell count decreased (Investigations) | 1 (5) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 3 (3) | 15 (17) | 13 (25) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 10 (12) | 1 (2) | 3 (3) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Open-label study with a small patient cohort, not designed for cross-arm efficacy comparison. Efficacy judged by investigator assessment with no BICR.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT03742102/Prot_002.pdf
  • Statistical Analysis Plan (2024-12-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT03742102/SAP_001.pdf